CLINICAL TRIAL: NCT06551545
Title: Tryptophan Metabolism in Healthy Young Adults in Response to Graded Tryptophan Intakes: a Pilot Study
Brief Title: Tryptophan Metabolism in Healthy Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Principal investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1000081438
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: adults; healthy; tryptophan; tryptophan breakdown; indicator amino acid oxidation; stable isotope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Tryptophan in healthy young adults (18-45 years) (Experimental): Tryptophan intake levels, up to 5 levels, will be tested in a random order in all subjects
  Interventions: Dietary Supplement: Tryptophan intake

INTERVENTIONS:
Dietary Supplement: Tryptophan intake — There are 5 different tryptophan test intake levels ranging from 2, 3, 4.5, 6, 8 mg.kg-1.day.1

SUMMARY:
Tryptophan is an essential amino acid needed for growth and bodily functions. It is used to make serotonin which is needed for the brain to develop and function properly. However, when the body is stressed, tryptophan is broken down into compounds that can cause harm to the brain. Premature babies who get nutrition through their vein [i.e. total parenteral nutrition (TPN)] can experience this type of stress. The amount of tryptophan in TPN solutions is much higher than what premature babies need and can produce too much harmful compounds. So, it is important to study the amount of these compounds made from tryptophan. But there are no methods available to study this. Therefore, the goal of this study is to develop a method to measure the compounds made from tryptophan breakdown in adults so that it can be used for preterm babies on TPN later.

DETAILED DESCRIPTION:
Tryptophan is an essential amino acid and must be obtained from the diet. In addition to its essential role in protein synthesis, tryptophan has diverse and complex physiological functions via various metabolic pathways. Two primary metabolic pathways include the kynurenine and serotonin pathways. Tryptophan is the only precursor for both the kynurenine and serotonin pathways. Since these two pathways share tryptophan as the common nitrogenous substrate, a competition between these pathways is demonstrated. This can result in serotonin deficiency when kynurenine pathway is activated and may contribute to the pathophysiology of developing neurological disease. Furthermore, metabolites of the kynurenine pathway can exert neurotoxic effects because they can cross the blood brain barrier to reach the central nervous system (CNS). Evidence thus far indicates that the contribution of the different pathways of tryptophan metabolism can differ based on the physiological and pathological status. However, there is no clear evidence of whether the kynurenine pathway takes precedence over synthesis of protein (for growth) or serotonin during immune activation. There are also no investigations examining the impact of tryptophan intake during immune activation, for the purposes of this study meaning any activity by the immune system, on the production of neurotoxic metabolites of the kynurenine pathway.

Tryptophan uptake from parenteral nutrition fed to preterm neonates with current amino acid solutions may be about 2-2.5 times the estimated requirement based on data from neonatal piglets. Long-term effects of this excess intake in this vulnerable population are unknown. The potential adverse effects of increased catabolism via the kynurenine pathway during stress on growth and neurodevelopment of hospitalized preterm infants has not been explored. A method to quantify the partitioning of tryptophan between the different pathways will be highly beneficial but has not been established in humans. This will enable studies in parenterally fed neonates to assess whether tryptophan concentrations in current commercial amino acid solutions produce toxic metabolites or serotonin deficiency, which can contribute to neurocognitive deficits seen in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. Aged 18 to 45 years old (inclusive)
3. In good general health as evidenced by medical history, physical health and biochemistry
4. Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine and CRP levels within normal ranges for age.

Exclusion Criteria:

1. Presence of chronic disease and/or acute illness known to affect protein/amino acid metabolism (e.g. HIV, diabetes, cancer, liver or kidney disease, neurological conditions including depression and anxiety, hypo- / hyperthyroidism, inflammatory conditions,, anemia, acute cold or flu)
2. Taking medications known to affect protein/AA metabolism (e.g. steroids, anti-inflammatory medications, acetaminophen, selective serotonin reuptake inhibitors (SSRI))
3. Inability to tolerate the diet (i.e. allergy)
4. Significant weight loss during the past month or consumption of weight reducing diets.
5. Significant caffeine consumption (>2 cups per day)
6. Significant consumption of alcohol (>1 drink per day i.e. 1 beer or ½ glass of wine).
7. Unwilling to have blood drawn from a venous access or using a ventilated hood indirect calorimeter for the purposes of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Fractional Synthesis Rate (FSR) of tryptophan metabolites | 10 hours
  Enrichment of L-[15N2]tryptophan and its metabolites (15N2-L-kynurenine, 15N-kynurenic acid, 15N-quinolinic acid, 15N2-serotonin and 15N-5-hydroxyindole acetic acid) in plasma and urine following orally administered tracer, L-[15N2]tryptophan.
Steady state | 10 hours
  Time at which plasma and urine enrichment of L-[15N2]tryptophan reaches steady-state.

SECONDARY OUTCOMES:
Partitioning of tryptophan metabolism | 10 hours
  Partitioning of tryptophan between kynurenine and serotonin pathway at tryptophan intake below and above requirements
Fractional synthesis rate (FSR) | 10 hours
  Fractional synthesis rate (FSR) of metabolites of tryptophan (15N2-L-kynurenine, 15N-kynurenic acid, 15N-quinolinic acid, 15N2-serotonin and 15N-5-hydroxyindole acetic acid) at isotopic steady state

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No